CLINICAL TRIAL: NCT02468115
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Antiviral Activity of a Single Intravenous Dose of VIS410 in Healthy Subjects After a Viral Inoculation With Influenza A (H1N1)
Brief Title: Influenza Challenge Study of VIS410 in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS410-201
Record Dates: First submitted 2015-06-01; First posted 2015-06-10 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — VIS410 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VIS410 (Experimental): Single intravenous fixed dose of VIS410
  Interventions: Drug: VIS410
- Placebo (Placebo Comparator): Single intravenous infusion of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIS410 — Single fixed IV dose of VIS410
  Arms: VIS410
Drug: Placebo — Single IV dose of placebo
  Arms: Placebo

SUMMARY:
A phase 2 a study to assess the safety profile and the effect of VIS410 in healthy subjects after inoculation with influenza A virus (H1N1).

DETAILED DESCRIPTION:
This is a phase 2a randomized, double-blind, placebo-controlled study to be conducted in healthy volunteers. The study is designed to compare an infusion of a single dose of VIS410 against placebo. Eligible volunteers will be admitted to the clinical center and will receive a single intranasal administration of influenza A (H1N1). One day (24h) after inoculation, subjects will receive a single administration of VIS410 or placebo. Subjects will be confined in the clinical center for 10 days after virus administration.

Assessment of safety will be determined from vital sign measurements, physical examinations, hematology, chemistry and urinalysis laboratory testing, 12-lead electrocardiograms (ECGs), pulmonary function, use of concomitant medications, and review of adverse events (AEs) should they occur. During confinement in the clinical center a symptom score card of influenza symptoms will be completed three times a day; nasopharyngeal swabs will be obtained three times a day and assayed for the presence of influenza virus and VIS410 concentration; serum samples will be assayed for VIS410 and the presence of cytokines. Upon release from the clinical center subjects will return for follow-up visits on days 14, 28 and either 56 or 84.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of age 18-45 years, inclusive, at the time of informed consent.
2. Women should fulfill one of the following criteria:

   * Post-menopausal; either amenorrhea ≥ 12 months or follicle stimulating hormone > 40 mIU/mL.
   * Surgically sterile; bilateral oophorectomy, hysterectomy, or tubal ligation.
   * Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception until the end of the study.
   * Must be sexually inactive by abstinence which is consistent with the preferred and usual lifestyle of the subject.
3. Women of childbearing potential must have a negative pregnancy test at screening (serum) and on Day -2 (urine).
4. Non-vasectomized (or vasectomized less than 6 months prior to dosing) male subjects must use an effective birth control method (see Inclusion Criterion 2).
5. Seronegative for the challenge virus (HAI ≤ 10).

Exclusion Criteria:

1. Known or suspected intolerance or hypersensitivity to the investigational study drug or virus.
2. Has an acute or chronic medical condition that would render the investigational study drug unsafe or would interfere with the evaluation of the responses.
3. Subjects receiving medications that affect the immune system.
4. Significant adulthood history of seasonal hay fever or a seasonal allergic rhinitis or perennial allergic rhinitis or chronic or nasal or sinus condition.
5. Subjects who have received any vaccination within the last 3 months or influenza vaccine within the last 6 months.
6. Subjects with a confirmed diagnosis of influenza A within the last 6 months prior to screening.
7. Subjects with abnormal nasal structure (including septal deviation and nasal polyps), chronic sinusitis, or reason (i.e., intolerance) that complicates nasopharyngeal swabbing.
8. Presence of lung disease, asthma, or chronic obstructive pulmonary disease.
9. Has a history of alcohol or drug abuse.
10. A positive HIV antibody screen, HBsAg, HBcAb or hepatitis C antibody screen.
11. Cancer or treatment for cancer, within 3 years, excluding basal cell carcinoma of the skin, which is allowed.
12. Presence of immunosuppression or any medical condition that may be associated with impaired immune responsiveness.
13. Anticipated presence of a household contact with potential immunosuppression.
14. History of Guillain-Barré syndrome.
15. Current professional activity as a healthcare worker who will return to work within 2 weeks following challenge.
16. Anticipated presence of a pregnant household contact, within 2 weeks following challenge.
17. Women who are pregnant or breast-feeding, or consider becoming pregnant.
18. Acute disease within 2 weeks prior to challenge.
19. Elevated white blood cell count above 10.90 x 109/L or an absolute neutrophil count above 7.5 x 109/L.
20. Current enrollment in any other investigational drug study or disease study or participation in an investigational drug study.
21. Any other reasons for which the investigator considers the subject unfit for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the effect of VIS410 on the area under the curve of viral shedding over time. | 56-84 days
  The viral AUC will be measured, qRT-PCR, and compared between treatment groups
To assess the safety profile of VIS410 | 56-84 days
  The proportion of subjects with post-infusion adverse events will be compared between treatment groups.

SECONDARY OUTCOMES:
Assess the effects of VIS410 on viral shedding | 10 days
  The peak viral load and time to cessation of shedding will be measured (qRT-PCR and TCID50)
Assess the pharmacokinetics of VIS410 in serum | 56-84 days
  The following PK parameters will be calculated: Cmax, tmax, AUC, t1/2, Vd, Cl
Assess the immunogenicity of VIS410 | 56-84 days
  The development of anti-drug antibodies will be measured
Assess the effect of VIS410 on clinical symptoms | 10 days
  The duration of symptoms will be compared between treatment groups
Assess antibody to challenge strain | 28 days
  The HAI antibody titer will be measured

OTHER OUTCOMES:
Assess the pharmacokinetics of VIS410 in the nasal mucosa | 10 days
  The following PK parameters will be calculated: Cmax, tmax, AUC, t1/2
Assess viral target sequence in viral isolates to determine emergence of resistant viruses | 28 days
  Sequencing will be used to determine the emergence of resistant virus in the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: M Petkova, Principal Investigator — SGS Life Sciences, a division of SGS Belgium NV
Locations (1):
- SGS Life Sciences, Antwerp, Belgium

REFERENCES:
- [Derived] Sloan SE, Szretter KJ, Sundaresh B, Narayan KM, Smith PF, Skurnik D, Bedard S, Trevejo JM, Oldach D, Shriver Z. Clinical and virological responses to a broad-spectrum human monoclonal antibody in an influenza virus challenge study. Antiviral Res. 2020 Dec;184:104763. doi: 10.1016/j.antiviral.2020.104763. Epub 2020 Mar 7. PMID 32151645